CLINICAL TRIAL: NCT00959426
Title: A Phase 1 Placebo-Controlled Trial To Assess The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Multiple Escalating Oral Doses Of PF-04620110 In Otherwise Healthy Overweight And Obese Adult Subjects
Brief Title: A Multiple Dose Study Of PF-04620110 In Overweight And Obese, Otherwise Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B0961002
Record Dates: First submitted 2009-08-12; First posted 2009-08-14 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Obesity; Overweight; Healthy
Keywords: - Mutliple Ascending Dose Study in Overweight Subjects - Body Weight - Signs and Symptoms
MeSH Terms: conditions — Obesity; Overweight | interventions — PF-04620110

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04620110 (Experimental)
  Interventions: Drug: PF-04620110
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04620110 — Multiple oral doses of PF-04620110 will be given. The specific dose will depend on the cohort to which the subject is assigned Initial planned doses are 1, 3, 5, 10 and 20 mg but may be modified based on emerging PK and safety data.
  Arms: PF-04620110
Drug: Placebo — Subjects will be given placebo or PF-04620110. Anticipated total daily doses for Cohorts A, B, C, D, E, F and G are 1, 3, 5, 10 and 20 mg. In each Cohort 9 subjects will receive active treatment and 3 will receive placebo for 14 days. Doses shown may be adjusted upwards or downwards and may be adjusted to include intermediate doses during the study based on ongoing safety, tolerability and PK results, but will not be projected to exceed established PK stopping criteria.
  Arms: Placebo Comparator

SUMMARY:
PF-04620110 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics, and pharmacodynamics, of multiple oral doses of PF-04620110.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years
* Body Mass Index (BMI) of 26.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To assess safety and tolerability of PF-04620110 will be assessed by physical examinations, adverse event monitoring, 12-lead ECGs, vital sign, andc linical safety laboratory measurements. | Baseline to 2 weeks
To characterize the PK of PF-04620110 following multiple oral doses in otherwise healthy overweight and obese subjects. | Baseline to 2 weeks
To characterize the effect of PF-04620110 on postprandial lipid metabolism measures. | Baseline to 2 weeks

SECONDARY OUTCOMES:
To examine additional pharmacodynamic markers in response to multiple oral doses of PF-04620110. | Day -1 and Day 14
Secondary Pharmacodynamic Endpoints in response to a liquid meal test | Day -1 and Day 14
Triglyceride excursions | Day -1, Day 1, and Day 14
Glucose, insulin, and C-peptide excursions | Day -1 and Day 14
Gut hormone excursions- including active GLP-1, total amide GLP-1, ghrelin, GIP, and PYY | Day -1 and Day 14
Additional Secondary Pharmacodynamic Endpoint: Fasting adiponectin | Day -1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Amin NB, Saxena AR, Somayaji V, Dullea R. Inhibition of Diacylglycerol Acyltransferase 2 Versus Diacylglycerol Acyltransferase 1: Potential Therapeutic Implications of Pharmacology. Clin Ther. 2023 Jan;45(1):55-70. doi: 10.1016/j.clinthera.2022.12.008. Epub 2023 Jan 21. PMID 36690550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961002&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-04620110%20In%20Overweight%20And%20Obese%2C%20Otherwise%20Healthy%20Volunteers